CLINICAL TRIAL: NCT06931873
Title: Neoadjuvant Radiochemotherapy Combined With QL1706 for MSS-type Low Rectal Cancer: a Prospective, Exploratory, Multicohort Study
Brief Title: Neoadjuvant Radiochemotherapy Combined With QL1706 for Low Rectal Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Director of Department of Colorectal Surgery, Changhai Hospital, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCRQ
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort1 (Experimental): Patients with low rectal cancer, clinical stage cT1-3N0M0
  Interventions: Combination Product: SCRT+Capoex+QL706
- Cohort2 (Experimental): Patients with low locally advanced rectal cancer with clinical stage cT4N0M0 or cTanyN+M0
  Interventions: Combination Product: LCRT+Capoex+QL706

INTERVENTIONS:
Combination Product: SCRT+Capoex+QL706 — Using a short-course radiotherapy treatment protocol, the primary tumor and high-risk areas were irradiated with a tumor dose of 25 Gy (5 Gy/treatment × 5 treatments); 2 weeks of rest after the end of radiotherapy were followed by 4 cycles of Capoex combined with QL706.
  Arms: Cohort1
Combination Product: LCRT+Capoex+QL706 — Using a long course radiotherapy treatment protocol, the primary tumor and high-risk areas were irradiated with a tumor dose of 50 Gy (2 Gy/treatment x 25 treatments); a 2-week break at the end of radiotherapy was followed by 4 cycles of Capoex combined with QL706.
  Arms: Cohort2

SUMMARY:
This study investigates the efficacy of neoadjuvant radiotherapy combined with QL1706 in MSS-type low-grade rectal cancer. This study is a prospective multicohort study, with cohort 1 intended to include patients with low grade early rectal cancer (cT1-3N0M0) and cohort 2 intended to include patients with low grade locally advanced rectal cancer (cT4N0M0 or cTanyN+M0). Each cohort included 30 subjects receiving neoadjuvant radiotherapy combined with QL1706 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to receive neoadjuvant therapy.
2. Aged 18-75 years, regardless of gender.
3. Diagnosed with low-lying rectal adenocarcinoma (tumor located ≤7 cm from the anal verge) via colonoscopy, endorectal ultrasound, and pelvic high-resolution MRI, without distant metastasis.
4. Histopathologically confirmed rectal adenocarcinoma.
5. Good patient compliance, able to attend follow-up visits as required.
6. ECOG performance status score of 0-1.
7. Laboratory tests meeting the following criteria:

   i. WBC ≥3.5×10^9/L, ANC ≥1.8×10^9/L, platelets ≥100×10^9/L, hemoglobin ≥100 g/L.

   ii. INR ≤1.5, APTT ≤1.5×ULN, or PTT ≤1.5×ULN. iii. Total bilirubin ≤1.25×ULN; ALT/AST ≤5×ULN. iv. 24-hour creatinine clearance ≥50 mL/min or serum creatinine ≤1.5×ULN.
8. Voluntary signed informed consent.

Exclusion Criteria:

1. History of malignant colorectal tumors.
2. Patients requiring emergency surgery (e.g., intestinal obstruction, perforation, or hemorrhage).
3. Known allergy to capecitabine, oxaliplatin, PD-L1 inhibitors, CTLA-4 inhibitors, or related drugs.
4. Histopathology indicating poorly differentiated adenocarcinoma or signet ring cell carcinoma.
5. Unstable systemic diseases, including but not limited to:

   Severe infection, uncontrolled diabetes, refractory hypertension, unstable angina, cerebrovascular accident, myocardial infarction, congestive heart failure, life-threatening arrhythmias, or severe hepatic/renal/metabolic disorders.
6. Conditions (e.g., psychiatric disorders, substance abuse) that may increase treatment risk, compromise compliance, or confound study results.
7. Participation in another interventional clinical trial or use of investigational drugs within 30 days prior to screening.
8. Pregnancy, lactation, or refusal to use effective contraception during the study.
9. Other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2035-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | After neoadjuvant therapy 1 month or after surgery 1 month
  Includes clinical complete response rate (cCR) and pathologic complete response rate (pCR)

SECONDARY OUTCOMES:
Overall survival | 3 years /5 years
  Overall survival
Disease Free survival | 3 years /5 years
  Disease Free survival
Wexner Fecal Incontinence Score (Wexner Score) | After neoadjuvant therapy 3 months or after surgery 3 months
  Evaluates the severity of fecal incontinence (frequency and type). Includes frequency of solid/liquid/gas incontinence, need for pad use, and impact on daily life. Total score ranges from 0-20; higher scores indicate more severe incontinence (0 = full control, 20 = complete incontinence).
Low Anterior Resection Syndrome Score (LARS Score) | After neoadjuvant therapy 3 months or after surgery 3 months
  Assesses bowel dysfunction (LARS syndrome) in patients after low anterior resection for rectal cancer. Includes abnormal bowel frequency, urgency/incontinence, fragmented defecation, and difficulty emptying the bowel. Total score ranges from 0-42, categorized as no LARS (0-20), minor LARS (21-29), or major LARS (≥30). Higher scores indicate worse symptoms; lower scores are better.
Short-Form 36 Health Survey (SF-36 Score ) | After neoadjuvant therapy 3 months or after surgery 3 months
  Broadly evaluates quality of life across eight domains: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain is scored 0-100; higher scores reflect better health in that domain. Higher total scores are better (100 = optimal health status).